CLINICAL TRIAL: NCT05278416
Title: Regular Home Use of Dual-light Photodynamic Therapy in the Management of Chronic Periodontitis.
Acronym: HOPE-CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koite Health Oy (Industry)
Collaborators: University of Helsinki (Other); Metropolia University of Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KHE2021Metro (HOPE-CP)
Record Dates: First submitted 2022-02-07; First posted 2022-03-14 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Periodontitis
Keywords: Lumoral; Lumorinse; Periodontitis; Anti-bacterial photodynamic therapy; aPDT; Plaque; aMMP-8
MeSH Terms: conditions — Periodontitis; Plaque, Amyloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lumoral treatment -device and Lumorinse tablets (Active Comparator): Subjects will receive detailed instructions for the use of Lumoral treatment -device and Lumorinse tablets. Subjects will be instructed to use the Lumoral treatment -device and follow the protocol once a day.
  Interventions: Device: Lumoral treatment -device and Lumorinse tablets
- Standard of Care (No Intervention): Subjects will receive oral hygiene instructions for the sonic toothbrushing and the use of interdental cleaning devices. They will not receive an additional intervention.

INTERVENTIONS:
Device: Lumoral treatment -device and Lumorinse tablets — Subjects will use Lumoral treatment -device and Lumorinse tablets daily as per protocol.
  Arms: Lumoral treatment -device and Lumorinse tablets

SUMMARY:
The study is a single site, randomized clinical trial designed to determine the efficacy of the Lumoral treatment in periodontitis patients.

DETAILED DESCRIPTION:
Lumoral treatment is a CE-marked medical device developed to provide a potent, targeted antibacterial action on dental plaque in a home environment. The device mechanism of action is antibacterial photodynamic therapy. The device is used by swishing a mouth rinse, strongly adhering to dental plaque. The plaque-adhered photoactive mouth rinse can be activated by a simple use light applicator. The antibacterial efficacy far exceeds chlorhexidine, without side effects in long-term use. Preliminary results have shown a promising anti-inflammatory response in addition to plaque reduction.

This early-stage study is designed to determine the efficacy of the Lumoral method in periodontitis patients. Improved supragingival plaque control can help to also sustain subgingival plaque management in the long term. In addition, the device might have a photobiomodulation effect on periodontal tissues.

ELIGIBILITY:
Inclusion Criteria:

* Periodontal disease stage I-III, according to criteria the American Academy of Periodontology (AAP) with at least 2 mm interdental CAL in the site of greatest loss
* Age of 18-85 years
* Presence of > 20 teeth
* Agreement to participate in the study and to sign a written consent form

Exclusion Criteria:

* Untreated/uncontrollable diabetes mellitus (DM) with HbA1c >7%, and HbA1c > 8 if insulin treated DM
* Any systemic disease (e.g., wound healing dysfunctions) that could alter the progression of periodontal disease
* Use of medicine that would affect the periodontal tissue within the last 6 months (antibiotics, anti-inflammatories, anticonvulsants, immunosuppressants, or calcium channel blockers, including doxycycline, bisphosphonates and chlorhexidine)
* Periodontal treatment during the previous 3 months
* Allergic to the photosensitizer
* Presence of major physical limitation or restriction that prohibit the hygiene procedures used in the study protocol
* Removable major prosthesis or major orthodontic appliance
* Active smoking, or habitual use of smokeless tobacco products
* Pregnancy or lactation
* A need for a hopeless teeth extraction, or open cavities in need for immediate endodontic treatment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2025-04-14 (Actual); Study Completion 2025-04-29 (Actual)

PRIMARY OUTCOMES:
Bleeding on Probing (BOP) | 6 months
  Clinical change concerning bleeding on probing change. A full-mouth assessment at six sites per tooth (mesiobuccal, buccal, distobuccal, mesiolingual, lingual, distolingual). Gingival bleeding is considered as positive if bleeding occurs within 15 seconds after gentle probing with a probe at the sulcus. Dichotomous scoring to each site of the tooth as bleeding "1 present" and "0 absent". BOP is reported as the percentage (%) of sites with positive findings. Calculation formula: number of bleeding sites/ 6 times number of teeth.

SECONDARY OUTCOMES:
Clinical Attachment Level (CAL) | 6 months
  Observation of clinical attachment level:
  A full-mouth assessment, measured at six sites per tooth. Assessed as the distance from the cementoenamel junction (CEJ) to the bottom of the periodontal pocket (mm). To calculate CAL, two measurements are needed:
  distance from the gingival margin to the CEJ and PPD; in recession: PPD + gingival margin to the CEJ; in tissue overgrowth: PPD - gingival margin to the CEJ.
Periodontal Pocket Depth (PPD) | 6 months
  A full-mouth assessment, measured at six sites per tooth. Assessed from the base of the pocket to the gingival margin (mm)
Device-related adverse events | 6 months
  Absence of device-related serious adverse events or any patterns of device-related adverse events graded as moderate
Inflammation marker aMMP-8 measurement | 6 months
  Change in aMMP8-measurement reflecting the reduction in periodontitis grade. The oral rinse fluid sample collection and the aMMP-8 marker analysis will be performed using Periosafe test (Dentognostics GmbH) according to the manufacturer's instructions.
Visual Plaque Index (VPI) | 6 months
  Assessment of six index teeth, measured at four sites per tooth
  Dichotomous scoring to each site of the tooth as plaque "1 present" and "0 absent" VPI reported as the percentage (%) of sites with plaque Calculation formula: number of sites with plaque/ 4 times number of teeth.
OHIP-14 | 6 months
  Patient related objectives: Oral-related quality of life measurement (OHIP-14) questionnaire.
Patient-related objective: PCS questionnaire | 6 months
  Measurements of internal motivation to dental hygiene by Perceived Competence Scale (PCS) questionnaire.
Patient-related objective: OSCA questionnaire | 6 months
  Measurements of internal motivation to dental hygiene by Oral Self-Care Assessment (OSCA) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Timo Sorsa, Professor, Principal Investigator — Univeristy of Helsinki; Tommi Pätilä, Docent, Study Director — Koite Health
Locations (1):
- Metropolia University of applied sciences, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No